A Prospective, Randomized
Study Comparing The Outcome
of Large-Diameter vs SmallDiameter Glenospheres in
Primary Reverse Shoulder
Arthroplasty Using the ReUnion
System

NCT# 02768597

November 17, 2016

Protocol title: A Prospective, Randomized Study Comparing The

Outcome of Large-Diameter vs Small-Diameter Glenospheres in Primary Reverse Shoulder Arthroplasty Using the ReUnion System

Principal Investigator: Dr. Mark Morrey MD

Co-Principal Investigator: Dr. Joaquin Sanchez-Sotelo MD PhD

Sub-Investigators: Mrs. Ashley Pountney PA-C

Mr. Jordan Becker PA-C

Investigator Address: Dr. Mark Morrey MD

Consultant and Professor of Orthopedic Surgery

Mayo Clinic

200 First Street SW Rochester MN 55905

## **Summary**

A prospective, randomized, blinded clinical trial is proposed to compare the outcome of primary reverse shoulder arthroplasty using the Stryker ReUnion system with implantation of either a 40 mm glenosphere or a 36 mm glenosphere, both with either a +2 mm or a +6 mm offset. The Stryker ReUnion is a shoulder arthroplasty system approved by the FDA.

Each shoulder will be assessed preoperatively, at 3 weeks, 3 months, one year and two years. The primary end-point will be range of motion at one year. Additional end-points will include dislocation, stress fractures of the acromion, metal ion levels in peripheral blood, neurovascular complications, radiographic notching, implant mechanical failure and revision surgery.

#### Introduction

Reverse shoulder arthroplasty has emerged as a very successful procedure for selected patients with severe degeneration of the glenohumeral joint and a deficient rotator cuff. All reverse systems incorporate various degrees of modularity to adapt size, length and other biomechanical parameters to each specific individual. One such parameter is the size of the glenosphere. Smaller glenospheres are easier to implant and seem to provide a good outcome with many reverse systems. Theoretically, a larger glenosphere could provide larger arcs of motion, decrease notching and increase soft-tissue tension. However, the effect of glenosphere size on motion and complications is largely unknown; to date, no study has specifically analyzed clinically the effect of sphere size on reverse outcome.

Modularity with use of multiple metal trunions and Morse tapers also creates concerns regarding metal ions in peripheral blood, a problem well identified in the field of total hip arthroplasty.

# Purpose

The purpose of this study is to compare the outcome of primary reverse shoulder arthroplasty using the Stryker ReUnion system with implantation of either a large (40 mm) or a small (36 mm) glenosphere, both with either a +2 mm or a +6 mm of lateral offset.

### **Materials and Methods**

## Study design

This will be a prospective, randomized, blind clinical trial. Physician's assistants will supervise the running of the study and evaluate all patients. Randomization will be provided through a password-protected computer program developed by Mayo Clinic Division of Biostatistics personnel and communicated to the surgical team for listing. Physician assistants will be blinded regarding glenosphere size at the time of follow-up evaluations.

The indications and contraindication as outlined in Stryker's labelling will be strictly followed. Off-label use of the device is prohibited.

## Inclusion and exclusion criteria

### Inclusions:

- Subjects willing to sign the informed consent
- Male and non-pregnant female subjects ages 50 90 at the time of surgery
- Subjects requiring a primary reverse total shoulder arthroplasty
- Subjects with the diagnosis of cuff-tear arthropathy (CTA), massive irreparable rotator cuff tear (MRCT) or osteoarthritis (OA) with marked posterior subluxation or bone loss

#### **Exclusions:**

- Inability to comply with follow-up requirements
- Subjects with inflammatory arthritis
- Subjects with proximal humerus fractures
- Subjects with sequels of trauma
- Subjects that are immunologically compromised
- Subjects with an active or suspected latent infection in or about the shoulder
- Need to add a tendon transfer
- Need for structural humeral bone graft
- Pregnant subjects

## Randomization

In order to assign patients to specific treatment groups in an unbiased manner, randomization will occur prior to surgery.

After the patient has met the inclusion criteria and given full informed consent, he/she will be assigned to the treatment group. The randomization will be stratified by variables with potential confounding effects on the outcomes of interest. Specifically, patients will be stratified by gender (male/female), age group (50-65/66-80/81+) and underlying diagnosis. Within each stratum, subjects will be assigned to one of the two treatment groups using a computerized dynamic allocation program as mentioned before.

## Sample size

The target sample size was estimated using shoulder range of motion as the primary outcome, and a 15° between-group difference as being a clinically meaningful difference. In a recent study of a cohort of patients undergoing primary RSA, Steen et al (Steen, ISES, 2015) reported the following means and standard deviations of postoperative shoulder flexion, abduction, and external rotation:  $153.3 \pm 32.7$ , 140.4 $\pm$  37.4, and 47.1  $\pm$  38.9, respectively. If similar variability is observed in the proposed study, a sample of 100 subjects in each of the two groups (200 total) will provide 80% power to detect a difference of at least 13.1° in shoulder flexion, 14.9° in abduction, and 15.5° in external rotation as being statistically significant (alpha = 0.05, two-sided). In order to protect against a potential subject attrition rate of up to 10% due to drop out or loss to follow-up, the target sample size of 100 in each of the two main groups (36mm glenosphere and 40 mm glenosphere) will be increased to 110 per group (220) total. Although the primary comparisons will be between the 36mm and 40mm study groups, subjects will be enrolled and randomized such that within each group, half of the subjects will have a +2mm offset, and half will have a +6mm offset. Thus there will be 55 subjects with a 36 + 2mm glenosphere, 55 subjects with a 36 + 6mm glenosphere, 55 subjects with a 40 + 2mm glenosphere, and 55 subjects with a 40 + 6 mm glenosphere.

## Surgical technique

All procedures will be performed by two shoulder arthroplasty surgeons: Drs. Mark Morrey MD and Joaquin Sanchez-Sotelo MD PhD. The surgeons will implant the prosthesis according to the standard surgical technique for this particular implant system. A biceps tenotomy and tenodesis will be performed in all patients. The subscapularis tendon will be repaired at the end of the procedure when possible. Patients will receive one preoperative dose and two postoperative doses of IV antibiotics separated by a 6-8 hour period. All patients will receive an interscalenic brachial plexus block for pain control unless medically contraindicated. A shoulder immobilizer will be placed in the operating room once the procedure is completed and used for three weeks.

## **Hospitalization**

Patients will be admitted to the hospital on the day of their surgery, unless medical problems dictate earlier admission. Hospitalization of 1 day is routine for these patients, although uncontrolled pain or medical complications could lead to a more prolonged admission.

## Physical therapy

Both treatment groups will undergo the same program of postoperative care and physical therapy. A shoulder immobilizer will be used for three weeks. Active and active-assisted motion exercises for the elbow, wrist and hand will be initiated on day 1. Shoulder active-assisted motion exercises will be initiated at week 3. Isometrics will be added at week 6. Therabands will be added at week 8.

## Data collection

## Operative data collected

- Surgical time
- Cuff status preimplantation
- Biceps status preimplantation
- Glenoid bone loss (photograph) preimplantation
- Increase in muscle strain as measured with ultrasound elastography in the conjoined and deltoid muscles
  - Implants used
  - Intraoperative motion
  - Subscapularis repair

### Clinical data collected

- Demographic data
- Pain (visual analogue scale)
- Subjective shoulder value
- Active and passive range of motion in elevation, external rotation and internal rotation
- Strength in abduction, external rotation, and internal rotation
- Pain along the biceps tendon
- Biceps cramping
- Speed test
- Neurovascular exam
- Oxford shoulder score
- Quick-DASH score
- ASES score
- Satisfaction (visual analogue scale)
- Muscle strain measured with ultrasound elastography

## Laboratory studies

- CBC, sedimentation rate and C-reactive protein
- Metal ion levels for chrome, cobalt and nickel

### Imaging studies

- Plain radiographs (AP in external rotation, axillary, whole humerus markers)
- In-growth xrays (only postoperatively)
- Preoperative CT-Scan
- CT-scan at one year postoperatively

## Radiographic analysis

Preoperative radiographs and CT scans will be measured for canal sizing, bone dimensions and bone loss.

Postoperative radiographs will be measured for length, offset and glenoid version. They will be analyzed for component fixation, glenoid notching, stress fractures of the acromion and screw position. Post-op CT at one year will be obtained.

### Visits

### #1. Preoperative visit

- Clinical evaluation
- Plain radiographs
- CT scan with three dimensional reconstruction
- Laboratory studies
- Muscle strain measured with ultrasound elastography

## #2. Intra-Operative

- Muscle strain measured with ultrasound elastography

## #3. First postoperative visit at 3 weeks

Plain radiographs

## #4. Visits at 3 mo, 1 yr, 2 yr, 5 yrs

- Clinical evaluation
- Plain radiographs + ingrowth radiographs
- Laboratory studies
- CT Scan (only at one year)
- Muscle strain measured with ultrasound elastography (only at one year)

# **Complications**

Any serious complication that occurs related to the device will be documented. If patients are lost to follow-up, it will be noted accordingly.

### Recruitment

The physician assistant or research coordinator will carry this out. The study will be described to the patient in detail, and a consent form clearly stating the background and reasoning, will be given to the patient. A consent form will be signed by the patient and a study person authorized to obtain consent. One copy will be given to the participant, a second copy will be scanned in the patient's electronic medical record, and the original consent will be kept in the patient's study folder.

## **Competency**

Study participants must be able to give informed consent.

## Gender and Racial/Ethnic Distribution

No gender or racial/ethnic group will be intentionally excluded from this study.

### Risks

Participation in this study, involving FDA-approved devices, poses no increased risk to patients undergoing reverse total shoulder arthroplasty surgery. Risk and complications of this procedure include infection, nerve injury, bleeding, blood clots, persistent pain, persistent stiffness, loosening, wear, osteolysis and other forms of mechanical failure.

# **Analysis and Intended Publications**

The primary outcome will be shoulder range of motion in elevation, external rotation, and internal rotation at 1 year post surgery. Additional outcomes will include strength, pain, speed test, Oxford Shoulder Score, ASES score, Quick-DASH score, and patient satisfaction. The analysis will focus on comparing the subjects randomized to the small glenosphere to the patients randomized to the large glenosphere, at 1 year. Additional comparisons will be performed to evaluate data collected at the 3-month, 2-year, and 5-year time points. Variables comprised of discrete data will be analyzed using chi-square tests or Fisher's exact tests (if low expected cell counts are observed). Continuous variables will be analyzed using two-sample t-tests or Wilcoxon rank sum tests, if necessary and appropriate. Two-factor models may be used to analyze the effect of study group and time since surgery simultaneously, including the evaluation of potential interactions between these two factors. Modeling tools may include ANOVA, logistic regression, or generalized linear models, as appropriate based on examination of the data distribution and structure. Furthermore, separate analyses may be undertaken on specific patient subsets,

including those with a primary diagnosis of OA, CTA, or MRTC. Other possible analyses may involve metal ion levels following RSA, correlation of sarcomere length (as measured with ultrasound elastography) with radiographic parameters, biceps symptoms, and screw location and length. All statistical tests will be two-sided and p-values less than 0.05 will be considered significant.

### <u>Budget</u>

### See enclosed documents

#### 1-75

- 1. Wright J, Potts C, Smyth MP, Ferrara L, Sperling JW, Throckmorton TW. A quantitative analysis of the effect of baseplate and glenosphere position on deltoid lengthening in reverse total shoulder arthroplasty. International journal of shoulder surgery. 2015 Apr-Jun;9(2):33-7.
- 2. Wiater BP, Koueiter DM, Maerz T, Moravek JE, Jr., Yonan S, Marcantonio DR, et al. Preoperative deltoid size and fatty infiltration of the deltoid and rotator cuff correlate to outcomes after reverse total shoulder arthroplasty. Clinical orthopaedics and related research. 2015 Feb;473(2):663-73.
- 3. Wiater BP, Baker EA, Salisbury MR, Koueiter DM, Baker KC, Nolan BM, et al. Elucidating trends in revision reverse total shoulder arthroplasty procedures: a retrieval study evaluating clinical, radiographic, and functional outcomes data. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul 23.
- 4. Werner BS, Daggett M, Carrillon Y, Walch G. Evaluation of lengthening in reverse shoulder arthroplasty comparing X-rays and computerised tomography. International orthopaedics. 2015 May 5.
- 5. Walker D, Matsuki K, Struk AM, Wright TW, Banks SA. Scapulohumeral rhythm in shoulders with reverse shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul:24(7):1129-34.
- 6. Wagner ER, Houdek MT, Elhassan BT, Sanchez-Sotelo J, Cofield RH, Sperling JW. What Are Risk Factors for Intraoperative Humerus Fractures During Revision Reverse Shoulder Arthroplasty and Do They Influence Outcomes? Clinical orthopaedics and related research. 2015 Oct;473(10):3228-34.
- 7. Venne G, Rasquinha BJ, Pichora D, Ellis RE, Bicknell R. Comparing conventional and computer-assisted surgery baseplate and screw placement in reverse shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul;24(7):1112-9.
- 8. Torrens C, Guirro P, Santana F. The minimal clinically important difference for function and strength in patients undergoing reverse shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Sep 26.
- 9. Teusink MJ, Pappou IP, Schwartz DG, Cottrell BJ, Frankle MA. Results of closed management of acute dislocation after reverse shoulder arthroplasty. Journal of

- shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Apr;24(4):621-7.
- 10. Tashjian RZ, Burks RT, Zhang Y, Henninger HB. Reverse total shoulder arthroplasty: a biomechanical evaluation of humeral and glenosphere hardware configuration. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Mar;24(3):e68-77.
- 11. Tashjian RZ. CORR Insights: Implant Design Variations in Reverse Total Shoulder Arthroplasty Influence the Required Deltoid Force and Resultant Joint Load. Clinical orthopaedics and related research. 2015 Sep 22.
- 12. Stephens SP, Paisley KC, Giveans MR, Wirth MA. The effect of proximal humeral bone loss on revision reverse total shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Oct;24(10):1519-26.
- 13. Stephens BF, Hebert CT, Azar FM, Mihalko WM, Throckmorton TW. Optimal baseplate rotational alignment for locking-screw fixation in reverse total shoulder arthroplasty: a three-dimensional computer-aided design study. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Sep;24(9):1367-71.
- 14. Steen BM, Cabezas AF, Santoni BG, Hussey MM, Cusick MC, Kumar AG, et al. Outcome and value of reverse shoulder arthroplasty for treatment of glenohumeral osteoarthritis: a matched cohort. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Sep;24(9):1433-41.
- 15. Smith SL, Li BL, Buniya A, Lin SH, Scholes SC, Johnson G, et al. In vitro wear testing of a contemporary design of reverse shoulder prosthesis. Journal of biomechanics. 2015 Sep 18;48(12):3072-9.
- 16. Shi LL, Cahill KE, Ek ET, Tompson JD, Higgins LD, Warner JJ. Latissimus Dorsi and Teres Major Transfer With Reverse Shoulder Arthroplasty Restores Active Motion and Reduces Pain for Posterosuperior Cuff Dysfunction. Clinical orthopaedics and related research. 2015 Oct;473(10):3212-7.
- 17. Samitier G, Alentorn-Geli E, Torrens C, Wright TW. Reverse shoulder arthroplasty. Part 1: Systematic review of clinical and functional outcomes. International journal of shoulder surgery. 2015 Jan-Mar;9(1):24-31.
- 18. Saier T, Cotic M, Kirchhoff C, Feucht MJ, Minzlaff P, Glanzmann MC, et al. Early results after modular non-cemented reverse total shoulder arthroplasty: a prospective single-centre study of 38 consecutive cases. Journal of orthopaedic science: official journal of the Japanese Orthopaedic Association. 2015 Sep;20(5):830-6.
- 19. Sabesan VJ, Lombardo DJ, Khan J, Wiater JM. Assessment of the optimal shoulder outcome score for reverse shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Oct;24(10):1653-9.
- 20. Sabesan V, Callanan M, Sharma V, Wiater JM. Assessment of scapular morphology and surgical technique as predictors of notching in reverse shoulder arthroplasty. American journal of orthopedics (Belle Mead, NJ). 2015 May;44(5):E148-52.

- 21. Padegimas EM, Maltenfort M, Lazarus MD, Ramsey ML, Williams GR, Namdari S. Future patient demand for shoulder arthroplasty by younger patients: national projections. Clinical orthopaedics and related research. 2015 Jun;473(6):1860-7.
- 22. North LR, Hetzler MA, Pickell M, Bryant JT, Deluzio KJ, Bicknell RT. Effect of implant geometry on range of motion in reverse shoulder arthroplasty assessed using glenohumeral separation distance. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Sep;24(9):1359-66.
- 23. Morris BJ, Haigler RE, O'Connor DP, Elkousy HA, Gartsman GM, Edwards TB. Outcomes of staged bilateral reverse shoulder arthroplasties for rotator cuff tear arthropathy. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Mar;24(3):474-81.
- 24. Matsoukis J, Billuart F, Houssam K, Dujardin F, Walch G. Conversion of total shoulder arthroplasty to reverse shoulder arthroplasty made possible by custom humeral adapter. Orthopaedics & traumatology, surgery & research: OTSR. 2015 Sep 8.
- 25. Maier MW, Zeifang F, Caspers M, Dreher T, Klotz MC, Rettig O, et al. Can reverse shoulder arthroplasty in post-traumatic revision surgery restore the ability to perform activities of daily living? Orthopaedics & traumatology, surgery & research: OTSR. 2015 Apr;101(2):191-6.
- 26. Li X, Dines JS, Warren RF, Craig EV, Dines DM. Inferior glenosphere placement reduces scapular notching in reverse total shoulder arthroplasty. Orthopedics. 2015 Feb;38(2):e88-93.
- 27. Langohr GD, Giles JW, Athwal GS, Johnson JA. The effect of glenosphere diameter in reverse shoulder arthroplasty on muscle force, joint load, and range of motion. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jun;24(6):972-9.
- 28. Ladermann A, Denard PJ, Boileau P, Farron A, Deransart P, Terrier A, et al. Effect of humeral stem design on humeral position and range of motion in reverse shoulder arthroplasty. International orthopaedics. 2015 Sep 18.
- 29. King JJ, Farmer KW, Struk AM, Wright TW. Uncemented versus cemented humeral stem fixation in reverse shoulder arthroplasty. International orthopaedics. 2015 Feb;39(2):291-8.
- 30. Kiet TK, Feeley BT, Naimark M, Gajiu T, Hall SL, Chung TT, et al. Outcomes after shoulder replacement: comparison between reverse and anatomic total shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Feb;24(2):179-85.
- 31. Katz D, Valenti P, Kany J, Elkholti K, Werthel JD. Does lateralisation of the centre of rotation in reverse shoulder arthroplasty avoid scapular notching? Clinical and radiological review of one hundred and forty cases with forty five months of follow-up. International orthopaedics. 2015 Sep 4.
- 32. Hussey MM, Hussey SE, Mighell MA. Reverse shoulder arthroplasty as a salvage procedure after failed internal fixation of fractures of the proximal humerus: outcomes and complications. The bone & joint journal. 2015 Jul;97-b(7):967-72.
- 33. Hettrich CM, Permeswaran VN, Goetz JE, Anderson DD. Mechanical tradeoffs associated with glenosphere lateralization in reverse shoulder arthroplasty. Journal

of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul 31.

- 34. Hattrup SJ, Waldrop R, Sanchez-Sotelo J. Reverse Total Shoulder Arthroplasty for Post-traumatic Sequelae. Journal of orthopaedic trauma. 2015 Jul 30.
- 35. Hartzler RU, Steen BM, Hussey MM, Cusick MC, Cottrell BJ, Clark RE, et al. Reverse shoulder arthroplasty for massive rotator cuff tear: risk factors for poor functional improvement. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul 11.
- 36. Hartel BP, Alta TD, Sewnath ME, Willems WJ. Difference in clinical outcome between total shoulder arthroplasty and reverse shoulder arthroplasty used in hemiarthroplasty revision surgery. International journal of shoulder surgery. 2015 Jul-Sep;9(3):69-73.
- 37. Guven MF, Aslan L, Botanlioglu H, Kaynak G, Kesmezacar H, Babacan M. Functional outcome of reverse shoulder tumor prosthesis in the treatment of proximal humerus tumors. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul 31.
- 38. Greiner S, Schmidt C, Herrmann S, Pauly S, Perka C. Clinical performance of lateralized versus non-lateralized reverse shoulder arthroplasty: a prospective randomized study. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Sep;24(9):1397-404.
- 39. Gilot G, Alvarez-Pinzon AM, Wright TW, Flurin PH, Krill M, Routman HD, et al. The incidence of radiographic aseptic loosening of the humeral component in reverse total shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Oct;24(10):1555-9.
- 40. Gillespie RJ, Garrigues GE, Chang ES, Namdari S, Williams GR, Jr. Surgical exposure for reverse total shoulder arthroplasty: differences in approaches and outcomes. The Orthopedic clinics of North America. 2015 Jan;46(1):49-56.
- 41. Giles JW, Langohr GD, Johnson JA, Athwal GS. Implant Design Variations in Reverse Total Shoulder Arthroplasty Influence the Required Deltoid Force and Resultant Joint Load. Clinical orthopaedics and related research. 2015 Nov;473(11):3615-26.
- 42. Garcia GH, Taylor SA, DePalma BJ, Mahony GT, Grawe BM, Nguyen J, et al. Patient Activity Levels After Reverse Total Shoulder Arthroplasty: What Are Patients Doing? The American journal of sports medicine. 2015 Aug 27.
- 43. Fortun CM, Streit JJ, Horton SA, Muh SJ, Gillespie RJ, Gobezie R. Scapular neck length and implications for reverse total shoulder arthroplasty: An anatomic study of 442 cadaveric specimens. International journal of shoulder surgery. 2015 Apr-Jun;9(2):38-42.
- 44. Formaini NT, Everding NG, Levy JC, Santoni BG, Nayak AN, Wilson C, et al. The effect of glenoid bone loss on reverse shoulder arthroplasty baseplate fixation. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul 8.
- 45. Fink Barnes LA, Grantham WJ, Meadows MC, Bigliani LU, Levine WN, Ahmad CS. Sports activity after reverse total shoulder arthroplasty with minimum 2-year follow-up. American journal of orthopedics (Belle Mead, NJ). 2015 Feb;44(2):68-72.

- 46. Ferreira LM, Knowles NK, Richmond DN, Athwal GS. Effectiveness of CT for the detection of glenoid bone graft resorption following reverse shoulder arthroplasty. Orthopaedics & traumatology, surgery & research: OTSR. 2015 Jun;101(4):427-30.
- 47. Erickson BJ, Frank RM, Harris JD, Mall N, Romeo AA. The influence of humeral head inclination in reverse total shoulder arthroplasty: a systematic review. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jun;24(6):988-93.
- 48. Dilisio MF, Miller LR, Siegel EJ, Higgins LD. Conversion to Reverse Shoulder Arthroplasty: Humeral Stem Retention Versus Revision. Orthopedics. 2015 Sep 1;38(9):e773-9.
- 49. Day JS, Paxton ES, Lau E, Gordon VA, Abboud JA, Williams GR. Use of reverse total shoulder arthroplasty in the Medicare population. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 May;24(5):766-72.
- 50. Cusick MC, Hussey MM, Steen BM, Hartzler RU, Clark RE, Cuff DJ, et al. Glenosphere dissociation after reverse shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul;24(7):1061-8.
- 51. Costantini O, Choi DS, Kontaxis A, Gulotta LV. The effects of progressive lateralization of the joint center of rotation of reverse total shoulder implants. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul;24(7):1120-8.
- 52. Carpenter S, Pinkas D, Newton MD, Kurdziel MD, Baker KC, Wiater JM. Wear rates of retentive versus nonretentive reverse total shoulder arthroplasty liners in an in vitro wear simulation. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Sep;24(9):1372-9.
- 53. Black EM, Roberts SM, Siegel E, Yannopoulos P, Higgins LD, Warner JJ. Failure after reverse total shoulder arthroplasty: what is the success of component revision? Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jul 7.
- 54. Berton A, Gulotta LV, Petrillo S, Florio P, Longo UG, Denaro V, et al. The effect of humeral version on teres minor muscle moment arm, length, and impingement in reverse shoulder arthroplasty during activities of daily living. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Apr;24(4):578-86.
- 55. Berliner JL, Regalado-Magdos A, Ma CB, Feeley BT. Biomechanics of reverse total shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Jan;24(1):150-60.
- 56. Berhouet J, Kontaxis A, Gulotta LV, Craig E, Warren R, Dines J, et al. Effects of the humeral tray component positioning for onlay reverse shoulder arthroplasty design: a biomechanical analysis. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Apr;24(4):569-77.
- 57. Athwal GS, MacDermid JC, Reddy KM, Marsh JP, Faber KJ, Drosdowech D. Does bony increased-offset reverse shoulder arthroplasty decrease scapular notching? Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2015 Mar;24(3):468-73.

- 58. Athwal GS, Faber KJ. Outcomes of reverse shoulder arthroplasty using a mini 25-mm glenoid baseplate. International orthopaedics. 2015 Aug 1.
- 59. Alentorn-Geli E, Samitier G, Torrens C, Wright TW. Reverse shoulder arthroplasty. Part 2: Systematic review of reoperations, revisions, problems, and complications. International journal of shoulder surgery. 2015 Apr-Jun;9(2):60-7.
- 60. Wiater JM, Moravek JE, Jr., Budge MD, Koueiter DM, Marcantonio D, Wiater BP. Clinical and radiographic results of cementless reverse total shoulder arthroplasty: a comparative study with 2 to 5 years of follow-up. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2014 Aug;23(8):1208-14.
- 61. Stevens CG, Struk AM, Wright TW. The functional impact of bilateral reverse total shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2014 Sep;23(9):1341-8.
- 62. Schwartz DG, Cottrell BJ, Teusink MJ, Clark RE, Downes KL, Tannenbaum RS, et al. Factors that predict postoperative motion in patients treated with reverse shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2014 Sep;23(9):1289-95.
- 63. Raiss P, Zeifang F, Pons-Villanueva J, Smithers CJ, Loew M, Walch G. Reverse arthroplasty for osteoarthritis and rotator cuff deficiency after previous surgery for recurrent anterior shoulder instability. International orthopaedics. 2014 Jul;38(7):1407-13.
- 64. Poon PC, Chou J, Young SW, Astley T. A comparison of concentric and eccentric glenospheres in reverse shoulder arthroplasty: a randomized controlled trial. The Journal of bone and joint surgery American volume. 2014 Aug 20;96(16):e138.
- 65. Pappou I, Virani NA, Clark R, Cottrell BJ, Frankle MA. Outcomes and Costs of Reverse Shoulder Arthroplasty in the Morbidly Obese: A Case Control Study. The Journal of bone and joint surgery American volume. 2014 Jul 16;96(14):1169-76.
- 66. Middleton C, Uri O, Phillips S, Barmpagiannis K, Higgs D, Falworth M, et al. A reverse shoulder arthroplasty with increased offset for the treatment of cuff-deficient shoulders with glenohumeral arthritis. The bone & joint journal. 2014 Jul;96-b(7):936-42.
- 67. Maier MW, Caspers M, Zeifang F, Dreher T, Klotz MC, Wolf SI, et al. How does reverse shoulder replacement change the range of motion in activities of daily living in patients with cuff tear arthropathy? A prospective optical 3D motion analysis study. Archives of orthopaedic and trauma surgery. 2014 Aug;134(8):1065-71.
- 68. Levy JC, Everding NG, Frankle MA, Keppler LJ. Accuracy of patient-specific guided glenoid baseplate positioning for reverse shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2014 Oct;23(10):1563-7.
- 69. Jiang JJ, Toor AS, Shi LL, Koh JL. Analysis of perioperative complications in patients after total shoulder arthroplasty and reverse total shoulder arthroplasty. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2014 Dec;23(12):1852-9.
- 70. Hoenecke HR, Jr., Flores-Hernandez C, D'Lima DD. Reverse total shoulder arthroplasty component center of rotation affects muscle function. Journal of shoulder and elbow surgery / American Shoulder and Elbow Surgeons [et al]. 2014 Aug;23(8):1128-35.

- 71. Hasan SS, Gordon MP, Ramsey JA, Levy MS. Reverse shoulder arthroplasty using an implant with a lateral center of rotation: outcomes, complications, and the influence of experience. American journal of orthopedics (Belle Mead, NJ). 2014 Sep;43(9):E194-9.
- 72. Giuseffi SA, Streubel P, Sperling J, Sanchez-Sotelo J. Short-stem uncemented primary reverse shoulder arthroplasty: clinical and radiological outcomes. The bone & joint journal. 2014 Apr;96-b(4):526-9.
- 73. Cabezas AF, Gutierrez S, Teusink MJ, Schwartz DG, Hartzler RU, Santoni BG, et al. Kinematic impact of size on the existing glenohumeral joint in patients undergoing reverse shoulder arthroplasty. Clinical biomechanics (Bristol, Avon). 2014 Jun;29(6):622-8.
- 74. Berhouet J, Garaud P, Slimane M, Nicot J, Banah J, Waynberger E, et al. Effect of scapular pillar anatomy on scapular impingement in adduction and rotation after reverse shoulder arthroplasty. Orthopaedics & traumatology, surgery & research: OTSR. 2014 Sep;100(5):495-502.
- 75. Alta TD, Veeger DH, de Toledo JM, Janssen TW, Willems WJ. Isokinetic strength differences between patients with primary reverse and total shoulder prostheses: muscle strength quantified with a dynamometer. Clinical biomechanics (Bristol, Avon). 2014 Nov;29(9):965-70.